CLINICAL TRIAL: NCT07017920
Title: The Relationship Among Vitamin Deficiency/Insufficiency, Vitamin Supplementation, and Hypertensive Disorders of Pregnancy
Brief Title: Vitamin D and Hypertensive Disorders of Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-073
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hypertensive Disorders of Pregnancy
Keywords: vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Standard OB care with no screening for vitamin D level. (No Intervention): Patients will receive standard OB care with no screening for vitamin D level.
- Arm 2: Vitamin D screening and supplementation if needed (Experimental): Patients will receive standard OB care and will have a vitamin D level drawn with their other prenatal labs during an OB visit. If vitamin D insufficiency (less than 30 ng/mL) or deficiency (less than 20 ng/mL) is detected, the patient will be prescribed and provided a supplementation of 2000 IU of vitamin D daily for the remainder of the pregnancy.
  Interventions: Diagnostic Test: Vitamin D Levels measurement

INTERVENTIONS:
Diagnostic Test: Vitamin D Levels measurement — Patient will have a vitamin D level drawn with their other prenatal labs during an OB visit. If vitamin D insufficiency (less than 30 ng/mL) or deficiency (less than 20 ng/mL) is detected, the patient will be prescribed and provided a supplementation of 2000 IU of vitamin D daily for the remainder of the pregnancy.
  Arms: Arm 2: Vitamin D screening and supplementation if needed

SUMMARY:
The purpose of this study is to further investigate the association between vitamin D deficiency/insufficiency and hypertensive disorders of pregnancy by studying the impact of screening for vitamin D deficiency and supplementation when low levels of vitamin D are detected. Screening for vitamin D deficiency (less than 20 ng/mL) and insufficiency (less than 30 ng/mL) may determine the need for additional supplementation, as most prenatal vitamins only contain 400 IU of vitamin D. The rates of hypertensive disorders of pregnancy amongst patients who received supplementation and maintained adequate vitamin D levels will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 18-45 years old
* Receiving care at outpatient OB office of TriHealth's Women's Services Comprehensive OB-GYN Team with a plan to deliver at Bethesda North Hospital

Exclusion Criteria:

* Non-English speaking
* Unable to provide consent to research study participation
* Diagnosis of preexisting renal disease
* Diagnoses of preexisting chronic hypertension
* Diagnosis of cardiovascular diseases
* Diagnosis of conditions limiting fat absorption
* Diagnosis of sarcoidosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 594 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypertensive disorders of pregnancy | During pregnancy, up to 9 months
  Was patient diagnosed with a hypertensive disorder of pregnancy (preeclampsia or GHTN) per clinician judgement based on ACOG guidelines

IPD SHARING:
Plan to Share IPD: Undecided